CLINICAL TRIAL: NCT06600568
Title: Identification of Targetable Vulnerabilities in Redox Homeostasis Pathways as a Novel Therapeutic Approach for Human T-cell Malignancies
Brief Title: Novel Therapeutic Approach for Human T-cell Malignancies
Status: Recruiting | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Istituto Nazionale Tumori IRCSS-Fondazione G.Pascale (Unknown)
Responsible Party: Sponsor
Other Study IDs: ROSinTALL
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: T-Cell Leukemia/Lymphoma, Adult
Keywords: T-cell lymphoblastic leukemias (T-ALL); T-cell non-Hodgkin's lymphomas (T-NHL); NK cell neoplasia; ROS; apoptosis
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Translation analysis — Novel strategies to selectively eliminate neoplastic T cells by modulating intracellular ROS levels.

SUMMARY:
This multicenter translational study, with prospective and retrospective samples, aims to identify new strategies to selectively eliminate neoplastic T cells by modulating intracellular ROS levels.

Interactions between drugs capable of activating the apoptotic process (e.g., Venetoclax) and drugs capable of altering ROS homeostasis (e.g., inhibitors of the enzyme glucose-6-phosphate dehydrogenase) will be examined.

The most promising compounds will be selected based on results obtained in vitro on cell lines and PDX already available in the laboratory, and then will be assayed ex vivo in cells obtained from patients with resistant/refractory T-cell neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pre- and post-thymic T-cell leukemia/lymphoma
* Patients of both sexes
* Age of patients older than 18 years
* Patient is willing to provide written and signed informed consent for participation in the study

Exclusion Criteria:

-Serious illness or medical condition that does not allow the patient to be managed according to standard treatment protocols, including uncontrolled active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to a maximum of 120 patients (both retrospective and prospective) are expected to be enrolled during the study period. Specifically, a maximum of 40 patients will be enrolled for each of the following diseases: T-cell lymphoblastic leukemias (T-ALL); T-cell non-Hodgkin lymphomas (T-NHL); NK-cell neoplasms. For retrospective peripheral blood samples, bone marrow aspirates, and lymph node biopsies, which are available at the centers involved in the study, patients will be contacted again to ask for consent regarding this project.
  No additional clinical procedures are specifically required by participation in the present study. In fact, samples will be obtained from the material left over from samples taken for clinical procedures.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | Through study completion, an average of 2 years
  Response of leukemic cells to treatments that remodulate redox state and apoptosis from a molecular point of view, ex vivo,through the development of a multidimensional approach aimed at reducing the chemoresistance of T neoplasms

SECONDARY OUTCOMES:
Secondary outcome | Through study completion, an average of 2 years
  Development of drug combinations that can selectively eliminate T-cell leukemia/lymphoma cells
Secondary outcome | Through study completion, an average of 2 years
  Analysis of DNA, RNA, protein, and circulating markers of alterations present at baseline in patient samples; profiles obtained will be correlated with response to drug treatments in order to identify biomarkers predictive of response to treatment.
Secondary outcome | Through study completion, an average of 2 years
  Analysis of the efficacy of new drug combinations in vivo through the generation of PDX-based experimental mouse models derived from patients with T-cell malignancies.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Nazionale Tumori Fondazione G.Pascale, Napoli
  - Istituto Oncologico Veneto, Padua

IPD SHARING:
Plan to Share IPD: No